CLINICAL TRIAL: NCT03097718
Title: Central Proprioceptive Processing and Postural Control in Individuals With and Without Recurrent Non-specific Low Back Pain
Brief Title: Central Proprioceptive Processing and Postural Control in LBP
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Collaborators: Agentschap voor Innovatie door Wetenschap en Technologie (Other)
Responsible Party: Principal Investigator, Simon Brumagne, Professor, KU Leuven
Other Study IDs: 2016_SBrumagne_PropriocProcess
Record Dates: First submitted 2017-01-26; First posted 2017-03-31 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-specific low back pain: Individuals with recurrent non-specific low back pain
- Healthy control subjects: Healthy individuals without low back pain

SUMMARY:
This project aims to elucidate neural correlates of proprioceptive deficits in patients with recurrent non-specific low back pain, by studying whether brain activation patterns during the processing of proprioceptive signals from the ankle muscles and lower back muscles are altered compared to healthy control subjects.

DETAILED DESCRIPTION:
Low back pain is a highly prevalent health condition, with a reported lifetime prevalence of up to 84% worldwide. Currently, it induces more disability than any other health condition, such as depression, diabetes, chronic obstructive pulmonary disease or other musculoskeletal disorders. Approximately 85% of all low back pain complaints are non-specific, meaning that the pain cannot be attributed to a recognizable specific pathology such as an infection or vertebral fracture. While many patients with low back pain recover within a month, a large number of patients report a recurrence within one year. Current treatment interventions often remain unsuccessful, which highlights the current lack of knowledge on the underlying mechanisms of non-specific low back pain.

Postural control deficits have been identified as a key factor in the development and recurrence of non-specific low back pain. To achieve optimal postural control, the central nervous system needs to process, integrate and weigh proprioceptive signals from different body regions (e.g. ankle muscles and lower back muscles) with vestibular and visual inputs. Several studies have shown that patients with non-specific low back pain have a decreased ability to optimally weigh proprioceptive signals during standing, which leads to reduced postural robustness compared to pain-free individuals. More specifically, patients with low back pain dominantly rely more on proprioceptive signals from the ankle muscles and are not able to up-weigh proprioceptive signals from the lower back muscles when needed. This might be due to an impaired central processing of proprioceptive signals. However, up to now no studies have investigated central proprioceptive processing in patients with recurrent non-specific low back pain.

Therefore, this project aims to elucidate whether patients with recurrent non-specific low back pain showed altered brain activation patterns during the processing of proprioceptive signals from the ankle muscles and lower back muscles compared to healthy controls, by applying local muscle vibration during functional magnetic resonance imaging (fMRI).

ELIGIBILITY:
Inclusion Criteria for individuals with recurrent non-specific low back pain:

* Age: 20 - 50 years old
* At least six months of low back pain with or without referred pain to the buttock or thigh
* At least three episodes of disabling low back pain
* A score of at least 14% on the Oswestry Disability Index
* Willing to sign the informed consent
* Meets specific criteria related to MRI-research

Inclusion Criteria for healthy individuals

* Age: 20 - 50 years old
* No history of low back pain
* A score of 0% on the Oswestry Disability Index
* Willing to sign the informed consent
* Meets specific criteria related to MRI-research

Exclusion Criteria for both groups:

* History of major trauma and/or major orthopedic surgery of the spine, the pelvis or the lower quadrant
* One of the following conditions: Parkinson's disease, multiple sclerosis, Stroke with sequelae
* Radicular symptoms
* Using strong opioid medication or antidepressants
* Neck pain
* Ankle problems

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Leuven and surrounding area
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-01; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Brain activation during the processing of proprioceptive signals originating in the ankle muscles and lumbar paraspinal muscles | One time point, immediately after inclusion in the study
  Brain activation during the processing of proprioceptive signals originating in the ankle muscles (soleus muscle) and lumbar paraspinal muscles (multifidus muscles) is studied by applying muscle vibration to these muscles during fMRI. The test subjects participate in one scanning session, during which three fMRI runs with ankle muscle vibration and three fMRI runs with lumbar paraspinal muscles vibration are made in alternating order. Each fMRI run consists of three conditions: 'muscle vibration at 60 Hz' that stimulates muscle proprioceptors and vibrotactile skin receptors, 'muscle vibration at 20 Hz' that stimulates vibrotactile skin receptors (serves as a control condition) and 'rest'. During each fMRI run, the two 'vibration' conditions are presented three times during 18s-long blocks. Each' vibration' block is followed by a 18s-long 'rest' block.
Proprioceptive use during postural control | One time point, immediately after inclusion in the study
  Mean center-of-pressure displacement in response to soleus muscle and/or multifidus muscle vibration (60 Hz, 0.5 mm) during upright standing on two support surfaces.
  Condition A: stable support surface:
  * Upright standing, vision occluded (20s) - bilateral soleus and multifidus muscle vibration (15s) - upright standing (20s)
  * Upright standing, vision occluded (20s) - bilateral soleus muscle vibration (15s) - upright standing (20s)
  * Upright standing, vision occluded (20s) - bilateral multifidus muscle vibration (15s) - upright standing (20s)
  Condition B: unstable support surface (Airex balance pad elite):
  * Upright standing, vision occluded (20s) - bilateral soleus and multifidus muscle vibration (15s) - upright standing (20s)
  * Upright standing, vision occluded (20s) - bilateral soleus muscle vibration (15s) - upright standing (20s)
  * Upright standing, vision occluded (20s) - bilateral multifidus muscle vibration (15s) - upright standing (20s)

CONTACTS AND LOCATIONS:
Locations (1):
- Katholieke Universiteit Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brumagne S, Janssens L, Janssens E, Goddyn L. Altered postural control in anticipation of postural instability in persons with recurrent low back pain. Gait Posture. 2008 Nov;28(4):657-62. doi: 10.1016/j.gaitpost.2008.04.015. Epub 2008 Jun 9. PMID 18541428
- [Background] Claeys K, Dankaerts W, Janssens L, Pijnenburg M, Goossens N, Brumagne S. Young individuals with a more ankle-steered proprioceptive control strategy may develop mild non-specific low back pain. J Electromyogr Kinesiol. 2015 Apr;25(2):329-38. doi: 10.1016/j.jelekin.2014.10.013. Epub 2014 Oct 31. PMID 25467548
- [Background] Claeys K, Brumagne S, Dankaerts W, Kiers H, Janssens L. Decreased variability in postural control strategies in young people with non-specific low back pain is associated with altered proprioceptive reweighting. Eur J Appl Physiol. 2011 Jan;111(1):115-23. doi: 10.1007/s00421-010-1637-x. Epub 2010 Sep 8. PMID 20824281
- [Background] Brumagne S, Janssens L, Knapen S, Claeys K, Suuden-Johanson E. Persons with recurrent low back pain exhibit a rigid postural control strategy. Eur Spine J. 2008 Sep;17(9):1177-84. doi: 10.1007/s00586-008-0709-7. Epub 2008 Jul 2. PMID 18594876